CLINICAL TRIAL: NCT05189587
Title: A Preliminary Clinical Trial for Efficacy of Non-invasive Home-based Transcranial Electrical Stimulation (TES) Therapy in Patients With Intractable Chronic Tinnitus
Brief Title: Home-based Transcranial Electrical Stimulation (TES) in Patients With Chronic Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Jin Song, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUBH_ENT_TES
Record Dates: First submitted 2021-11-24; First posted 2022-01-12 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Tinnitus; Depression; Depressive Disorder; Hearing Disorders; Otorhinolaryngologic Diseases
Keywords: Transcranial electrical stimulation; Tinnitus
MeSH Terms: conditions — Tinnitus; Depression; Depressive Disorder; Hearing Disorders; Otorhinolaryngologic Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TES group (Experimental): Intervention: Device (transcranial electrical stimulation, TES)
  Interventions: Device: transcranial electrical stimulation (TES)
- sham TES group (Sham Comparator): Intervention: Device (transcranial electrical stimulation, TES)
  Interventions: Device: transcranial electrical stimulation (TES)
- Control group (No Intervention): Intervention: none

INTERVENTIONS:
Device: transcranial electrical stimulation (TES) — Transcranial electrical stimulation (tES) is a noninvasive brain stimulation technique that passes an electrical current through the cortex of the brain to alter brain function. The electrical current is applied to an individual's scalp usually via two or more electrodes, and whilst a large amount of the current is conducted between electrodes through soft tissue and skull (Vöröslakos et al. 2018), a portion of the current penetrates the scalp and is conducted through the brain, where it can alter neuronal excitability. By altering the activity of brain regions involved with a behaviour of interest, investigators can observe the resulting behavioral changes and so establish a causal link between the two (Reed et al. 2018).
  Arms: TES group; sham TES group

SUMMARY:
The investigators applied home-based transcranial electrical stimulation (TES) for neuromodulative treatment in patients with intractable chronic tinnitus.

DETAILED DESCRIPTION:
For treatment of motor and psychiatric disorders, transcranial electrical stimulation including transcranial direct current stimulation (tDCS), transcranial magnetic stimulation (TMS), or transcranial random noise stimulation (tRNS) are in use worldwidely. The investigators applied these neuromodulation techniques into patients with intractable chronic tinnitus for symptom relief. Experimental groups with 60 subjective tinnitus subjects will be consisted of three different treatment groups which are: TES group, TES with sham stimulation group, and control group. Subjects will be given 1.0 milliampere (mA) TES on bifrontal areas for neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

* Research volunteers with intractable chronic tinnitus who agreed to participate in the clinical trial were gathered from the tinnitus clinic of the Department of Otorhinolaryngology Head-and-Neck Surgery, Seoul National University Bundang Hospital

Exclusion Criteria:

* psychoactive drug user
* implanted material
* pacemaker user

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Tinnitus handicap inventory (THI) | the same 1 week after treatment
  The THI consists of 25 items, each with the 3 response options-yes (4 points), sometimes (2 points), and no (0 points)-resulting in a total score range from 0 to 100. A higher score denotes a higher tinnitus-related handicap.

SECONDARY OUTCOMES:
resting-state quantitative electroencephalography (rs-qEEG) | the same 1 week after treatment
  EEG activities in certain cortical regions within all 8 frequency bands will be compared. Specifically, as for the source localization analysis, standardized low-resolution brain electromagnetic tomography (sLORETA) will be employed to estimate the scalp-recorded electrical activity in each of the eight frequency bands (i.e., intracerebral sources). We will identify the cortical sources that generate the activities recorded by the scalp electrodes in each of the following eight frequency bands: delta (2-3.5Hz), theta (4-7.5Hz), alpha 1 (8-10Hz), alpha 2 (10-12Hz), beta 1 (13-18Hz), beta 2 (18.5-21Hz), beta 3 (21.5-30Hz), and gamma (30.5-44Hz). sLORETA computes neuronal electrical activity as current density (A/m2) without assuming a predefined number of active sources.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae EB, Lee JH, Song JJ. Single-Session of Combined tDCS-TMS May Increase Therapeutic Effects in Subjects With Tinnitus. Front Neurol. 2020 Mar 27;11:160. doi: 10.3389/fneur.2020.00160. eCollection 2020. PMID 32292383